CLINICAL TRIAL: NCT01747057
Title: Monitoring Resuscitation in Severe Sepsis and Septic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Antonio Artigas Raventós, Director of Critical Care Area, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MORESS
Record Dates: First submitted 2012-11-29; First posted 2012-12-11 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Hemodynamics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dynamic guide resuscitation (Experimental): This arm follows a resuscitation protocol based on dynamic-parameters-guided fluid management.
  Interventions: Behavioral: Dynamic-parameters-guided fluid management
- Standard resuscitation (Active Comparator): This arm follows a common resuscitation protocol based on Surviving Sepsis Campaign recommendations.
  Interventions: Behavioral: Standard-guided-fluid management

INTERVENTIONS:
Behavioral: Dynamic-parameters-guided fluid management — ● In preload-responsive patients defined by the following dynamic parameters: Patients fully adapted to mechanical ventilation* and with sinus rhythm.
  1. PPV >12%. PPV: Pulse pressure variation PPV = (PPmax-PPmin)/ [(PPmax+PPmin)/2] x100 (during 5 respiratory cycles)
  2. SVV > 12% (15). SVV: Stroke volume variation
     * A tidal volume (Vt) ≥ 7-10cc/kg in mechanically ventilated (in a controlled mode - control volume or control pressure) and well-adapted patients without any inspiratory effort should be guaranteed.
  Fluid loading must be performed with crystalloids (1omL/Kg) or colloids (5ml/Kg) every 30 minutes until PPV-SVV < 12%, while hypoperfusion signs are present. Continue resuscitation following Surviving Sepsis Campaign rules excluding more fluid administration (as described in the standard intervention once CVP>12).
  ● Non-preload responsive patients (defined as PPV or SVV < 12%) will resume the same protocol as responders when fluid response parameters are negative.
  Arms: Dynamic guide resuscitation
Behavioral: Standard-guided-fluid management — Fluid loading in patients with hypotension or elevated lactates until normalization of MAP (> 65mmHg) or CVP > 12mmHg. If CVP reaches > 12 mmHg and MAP remains < 65mmHg, norepinephrine should be started to reach MAP > 65mmHg. Once MAP is restored, if hypoperfusion signs persist (elevated lactate or urine output < 0.5mL/Kg/h), ScvO2/SvO2 must be measured. In order to reach a ScvO2 ≥70% or SVO2 ≥65%, consider giving blood transfusion if hemoglobin level (Hb) ≤ 7g/dL, and also consider dobutamine (initial dose 2,5 µg/kg/min, increased by 2,5 µg/kg/min every 30 min up to a maximum dose of 20 µg/kg/min, presence of arrhythmia, or FC>110bpm). At that point, if hypoperfusion signs remain present, consider restart protocol from the beginning.
  Arms: Standard resuscitation

SUMMARY:
Our hypothesis is that hemodynamic fluid resuscitation guided by dynamic parameters will improve outcome in patients with severe sepsis and septic shock, by limiting the deleterious effects of fluid overload.

DETAILED DESCRIPTION:
To evaluate the efficacy of dynamic parameters versus static measures to guide fluid resuscitation we pretend to detect a 10% relative reduction in mortality. In addition, we pretend to observe an improvement on the length of resuscitation time, mechanical ventilation and vasopressor support-free days, ICU and hospital length of stay, organ failure and renal function.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Clinical evidence of sepsis (microbiology confirmation, radiological or direct view - pus in biological fluid or surgical direct view-).
* ≥ 2 SIRS criteria:

  * Temperature < 36.0°C or > 38.0°C
  * Heart rate > 90 bpm
  * Respiratory rate > 20 rpm or PaCO2 < 32 mmHg or need of mechanical ventilation.
  * Leukocytes > 12.0 x109/L or < 4.0 x109/L
* Hemodynamic insufficiency defined as (at least one of the following):

  * Sustained systemic hypotension (systolic arterial pressure ≤ 90 mmHg or MAP < 65 mmHg) or a decrease in MAP of > 30 mm Hg in a hypertensive patient.
  * Need of vasopressors.
  * Tachycardia (HR > 110 bpm) or bradycardia (HR < 55 bpm)
  * Acute onset of oliguria, defined as a decreased urine output < 0.5 ml/kg/hr for ≥ 2 hours
  * Serum lactate > 2 mmol/l
  * Peripheral cyanosis, mottled skin, prolonged capillary refill
* Mechanical ventilation without any kind of inspiratory effort and Vt 7-10 mL/Kg, Pplateau < 30 mmH2O. Those patients with ARDS under mechanical ventilation will need to tolerate a tidal volume of at least 7 mL/Kg during 30 seconds while the plateau pressure remains < 30 mmH2O.
* Prior hemodynamic monitoring by arterial catheter.
* Central venous catheter.

Exclusion Criteria:

* Acute myocardial infarction < 7 days.
* Pregnancy
* Prior request of limited code status or expected life length lower than 3 months.
* Shock > 12h
* Cardiac arrhythmia
* Aortic valvular disease
* Inability to properly measure arterial pressure wave forms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 952 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-02 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Mortality at 28 days | 28 days after hospital admission

SECONDARY OUTCOMES:
Length of resuscitation | 72 hours after protocol inclusion
  * Vasopressor use and fluid load between 0h to 6h
  * Vasopressor use and fluid load between 7h to 72h
Ventilator-free days | 28 days after admission
  From 1 to 28 days over 28 days in a month.
Vasopressor-free days | 28 days after admission
  From 1 to 28 days over 28 days in a month.
Organ failure-free days | 28 days after admission
  Cardiovascular, CNS, renal, hepatic, coagulation abnormalities. From 1 to 28 days over 28 days in a month.
ICU length of stay | At ICU discharge (expected average 30 days after admission)
Hospital length of stay | At hospital discharge (expected average 45 days after hospital admission)
Renal function evolution | 3 days after study enrollment
  Creatinin clearance will be calculated every day for the first 3 days (Cockroft-Gault formula).
Mortality at 3 months | 3 months after admission

CONTACTS AND LOCATIONS:
Locations (1):
- Area de Critics. Hospital de Sabadell, Sabadell, Barcelona, Spain